CLINICAL TRIAL: NCT02689024
Title: A Multicenter Randomized Controlled Trial in Elderly Patients With Hip Fractures Comparing Continuous Fascia Iliaca Compartment Block to Systemic Opioids and Its Effect on Delirium Occurrence
Brief Title: Delirium in Elderly Patients With Trauma of the Hip
Acronym: DEPTHip
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment too slow; intervention was standard care in patients who were not included; acute care pathways changed due to policy regarding hip fracture patients
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Milan Ridderikhof, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL54580.018.15; 2015-003650-40 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-23 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Hip Fractures; Anesthesia
Keywords: Nerve block; Analgesia
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — Bupivacaine; Acetaminophen; Diclofenac; Ibuprofen; Naproxen; Dipyrone; Fentanyl; Morphine; Levobupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous FICB with local anesthetics (Experimental): With ultrasound guidance, a Fascia Iliaca Compartment Block will be administered and a catheter left in the compartment underneath the iliac fascia. This catheter will remain in place until two days after surgery.
  Initial pain treatment in the Emergency Department will be with 40 mL bupivacaine 0.25% or equipotent dosages of levobupivacaine or ropivacaine. Thereafter, until removal of the catheter, pain is treated by titrating local anesthetics according to pain scores.
  Interventions: Drug: Bupivacaine; Drug: Levobupivacaine; Drug: Ropivacaine
- Traditional care with systemic analgesia (Active Comparator): Traditional care (usual care) will be on the discretion of the treating physician or hospital protocols and will comprise of systemic opioids such as fentanyl or morphine.
  Usually, these opioids are combined with several other drugs, such as: paracetamol, NSAIDs (diclofenac or ibuprofen or naproxen) or dipyrone. (Inter)national guidelines advice morphine as first line agent in elderly patients with hip fractures, as longer acting analgesics are usually required.
  Interventions: Drug: Acetaminophen; Drug: Diclofenac; Drug: Ibuprofen; Drug: Naproxen; Drug: Dipyrone; Drug: Fentanyl; Drug: Morphine

INTERVENTIONS:
Drug: Bupivacaine — Local anesthetic: amide group ATC code N01BB01
  Other Names: Marcaine
  Arms: Continuous FICB with local anesthetics
Drug: Acetaminophen — Analgesic drug: Acetanilide derivate with analgetic and antipyretic properties ATC code N02BE01
  Other Names: Paracetamol
  Arms: Traditional care with systemic analgesia
Drug: Diclofenac — Non-Steroidal Anti-Inflammatory Drug: Acetic acid derivative ATC code M01AB05 Usual dosage is 50 mg t.i.d. orally or 75 mg b.i.d. intramuscularly. In the Netherlands, intravenous administration is not used.
  Arms: Traditional care with systemic analgesia
Drug: Ibuprofen — Non-Steroidal Anti-Inflammatory Drug: Propionic acid derivative ATC code M01AE01 Usual dosage is 400 mg t.i.d. or q.i.d. orally.
  Arms: Traditional care with systemic analgesia
Drug: Naproxen — Non-Steroidal Anti-Inflammatory Drug: Propionic acid derivative ATC code M01AE02 Usual dosage is initially 500 mg orally, followed by 250 mg b.i.d. or t.i.d.
  Arms: Traditional care with systemic analgesia
Drug: Dipyrone — Analgesic drug: Pyrazolone derivate with analgetic, antipyretic and antiphlogistic properties ATC N02BB02 Usual dosage is 1000 mg t.i.d. or q.i.d. orally and intravenously
  Other Names: Metamizole, Novalgin
  Arms: Traditional care with systemic analgesia
Drug: Fentanyl — Opioids: Phenylpiperidine derivative. Short-acting opioid. ATC code N02AB03 Usual dosage is 1 ug/kg intravenously and titrated guided by pain scores and possible side effects. Above the age of 60, dosages are usually divided in two in order to prevent adverse events.
  Arms: Traditional care with systemic analgesia
Drug: Morphine — Opioids: Natural opium alkaloid. Longer-acting opioid. ATC code N02AA01 Usual dosage is 0.1 mg intravenously and titrated guided by pain and possible side effects. Above the age of 60, dosages are usually divided in two in order to prevent adverse events.
  Arms: Traditional care with systemic analgesia
Drug: Levobupivacaine — Local anesthetic: amide group ATC code N01BB10
  Other Names: Chirocaine
  Arms: Continuous FICB with local anesthetics
Drug: Ropivacaine — Local anesthetic: amide group ATC code N01BB09
  Other Names: Naropin
  Arms: Continuous FICB with local anesthetics

SUMMARY:
A broken hip occurs frequently in elderly patients and is often very painful. Side effects of inadequately treated pain as well as the traditional drugs (administered through intravenous catheter) used to treat pain are, among others, a confusional state, called delirium. When pain medication is administered locally, only around the hip joint, pain might be treated more effectively and these side effects could be prevented. This is called a nerve block.

The current study evaluates the use of a continuous nerve block throughout the complete hospital admission with a catheter around the hip joint versus the use of traditionally used pain medication administered though an intravenous catheter in elderly patients with a broken hip. Half of all patients will receive the nerve block while in the emergency department and the other half will receive pain medication through the intravenous access.

DETAILED DESCRIPTION:
BACKGROUND Hip fractures occur frequently and are usually very painful. Pain itself is an indicator for increased risk of complications. A significant complication is delirium, occurring in up to 25% of all elderly patients with hip fractures. For a large proportion, triggers for development of delirium reaches back to the preoperative phase, where polypharmacy (including opioid use) and inadequately treated pain are major risk factors. Delirium is associated with negative health consequences, increased hospital stay, falls, higher mortality, decreased physical and cognitive function, re-hospitalization, increased risk of dementia and increased societal costs. Therefore, pain should be optimally treated as soon as possible, however the elderly patient poses a challenge in good pain treatment, because of physiological age-related changes, different drug effects, distribution, metabolism and elimination. Opioids frequently lead to respiratory depression, hypotension, nausea/vomiting and sedation in this vulnerable patient group. As a consequence, these drugs are often under dosed and pain treated insufficiently. Besides, drugs as opioids and NSAIDs have been associated with an increased delirium risk. A nerve block could alleviate these clinical issues.

An example of a nerve block frequently utilized in the Emergency Department (ED) is a Fascia Iliaca Compartment Block (FICB), in which local anesthetics are injected underneath the pelvic iliac fascia in order to block femoral, obturator and lateral cutaneous nerves to provide anesthesia of hip, thigh and knee. Case-series and historically controlled cohort studies show a single-shot FICB is a rapid, safe and easy procedure providing excellent analgesia, decreased opioid need and little risk of complications. Delirium as outcome was reported in one RCT; a decreased delirium incidence after using repetitive, blind, single-shot FICBs (not in the acute setting) with pethidine (with increased intrinsic risk of developing delirium) as comparison. In order to prevent the need for repetitive insertions, leaving a catheter would create a route in order to provide continuous analgesia with local anesthetics. Two case series describe this continuous FICB in hip fractures and reported good pain control and decreased length of hospital stay without any infectious complications. No comparison studies have been done with a continuous FICB.

The objective of the current study is to investigate whether the use of a continuous FICB, started early (in the ED) and continued throughout the complete clinical course of a hip fracture, will decrease occurrence of delirium in elderly patients with hip fractures.

METHODS This study is designed as a prospective, open, multi-center, randomized interventional trial. Patients will be allocated to continuous FICB or care as usual (according to national guidelines) in a 1:1 ratio and followed up until three months after hospital discharge.

SAMPLE SIZE AND DATA ANALYSIS The primary outcome (occurrence of delirium) is expected to be distributed normally. Although evidence to prevent delirium is scarce, an absolute reduction of 13% incidence has been reported previously after an intervention. The estimated delirium incidence according to literature is 25%. The hypothesis is that by using a continuous FICB administered very early in the clinical course in the ED, the incidence can be decreased from 25 to 12%. Superiority of the FICB versus usual care will be tested using the Chi Square Test. In order to detect a clinically relevant between-group-difference of 13% decrease in incidence, a significance level of 0.05 and 80% power will be used. For this analysis, each group will have 154 patients. When accounting for 10% loss to follow-up after three months, a total study population of 340 will be needed.

The primary analysis will be based on the intention to treat principle. Per protocol analysis will be performed to check robustness of results. Baseline characteristics will be presented using descriptive statistics. Ordinal data will be analyzed using Chi Square Test or Fisher exact test. Continuous data will be assessed by a Student's t-test if normally distributed or Mann Whitney U test if otherwise. Missing data will be corrected by multiple imputation.

An economic evaluation will be performed focusing on possible gained benefits of pain management with a continuous FICB compared to care as usual and the related health care costs. The economic evaluation will be performed from a societal perspective with a time horizon of three months and capturing the value of all resources utilized. The economic evaluation will be set up as a Cost-Effectiveness Analysis (CEA). Besides a CEA, a Budget Impact Analysis (BIA) will be performed according to the ISPOR Task Force principles.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged ≥ 55 years with
* a radiographically confirmed hip fracture

Exclusion Criteria:

* multiple injuries (polytrauma patients)
* previous adverse reaction or known allergy to local anaesthetics or opioids or paracetamol
* skin infection in proximity of injection site
* delirious state at presentation in the ED

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
occurrence of delirium | three months
  Diagnosis will be based on DSM-IV criteria. During hospital admission screening is actively. After discharge, information is gathered by contacting patients and family members, general practitioners or nursing facilities

SECONDARY OUTCOMES:
duration of delirium | three months
  duration is defined as the total number of days with delirium.
severity of delirium | three months
  severity is defined as percentage of patients with delirium duration > 2 days.
NRS pain scores | from hospital admission until 48 hours after surgery
  NRS pain scores during complete hospital stay, NRS pain scores will be recorded in the Emergency Department before the intervention as well as after the intervention at 30-minutes time intervals (this is according standard protocol in case opioids are administered). During hospital stay, during each nursing shift, a minimum of one NRS pain score is documented.
need for additional analgesia | hospital admission until 48 hours after surgery
  need for rescue analgesia will be documented during complete Emergency Department and hospital stay.
patient satisfaction | from hospital admission until 48 hours after surgery
  satisfaction of patients and health care staff regarding efficacy of pain treatment and method of pain treatment is recorded in the Emergency Department and daily during hospital admission (5-point Likert scales and reference questions).
length of hospital stay | from hospital admission until discharge; an average of 9 days
  defined as total consecutive days admitted in the hospital.
ICU admission | from hospital admission until discharge; an average of 9 days
  binary endpoint, whether patient is admitted to the ICU at any moment during hospital stay.
ICU length of stay | from hospital admission until discharge; an average of 9 days
  defined as total days admitted to the ICU department.
hospital re-admission rate | three months
  a re-admission occurs when a patient is admitted to the hospital within three months after initial discharge (from hip fracture related admission).
medical complications | three months
  all events regarding infections, renal- or pulmonary function and cardiovascular events will be accounted for.
surgical complications | three months
  defined as dislocations and fractures.
mortality | three months
  all cause in-hospital-mortality and mortality after hospital discharge.
activities of daily living | three months
  15-item modified Katz Index of Activities of Daily Living at three months after discharge. Baseline will be 2 weeks before presentation.
generic quality of life | three months
  generic HRQol (Euroqol - EQ-5D-5L) at three months after discharge. Baseline will be 2 weeks before presentation.
Oxford hip score | three months
  Oxford Hip Score after 3 months.
cognitive function with Mini Mental State Examination | three months
  Mini Mental State Examination at inclusion in the study, at hospital discharge and at three months after discharge.
cost effectiveness analysis | three months
  primary focus on direct medical costs, direct non-medical costs, indirect costs and productivity loss.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hollmann, MD, PhD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (5):
- Netherlands (5):
  - Tergooi Ziekenhuis, Hilversum, North Holland
  - Meander Medical Center, Amersfoort
  - Slotervaart Medical Center, Amsterdam
  - VU Medical Center, Amsterdam
  - Academic Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
After an embargo period data can be shared, depending on research question, objectives, statistics and methodology.

REFERENCES:
- [Background] Abou-Setta AM, Beaupre LA, Rashiq S, Dryden DM, Hamm MP, Sadowski CA, Menon MR, Majumdar SR, Wilson DM, Karkhaneh M, Mousavi SS, Wong K, Tjosvold L, Jones CA. Comparative effectiveness of pain management interventions for hip fracture: a systematic review. Ann Intern Med. 2011 Aug 16;155(4):234-45. doi: 10.7326/0003-4819-155-4-201108160-00346. PMID 21844549
- [Background] Bruce AJ, Ritchie CW, Blizard R, Lai R, Raven P. The incidence of delirium associated with orthopedic surgery: a meta-analytic review. Int Psychogeriatr. 2007 Apr;19(2):197-214. doi: 10.1017/S104161020600425X. Epub 2006 Sep 14. PMID 16973101
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] McCusker J, Cole MG, Dendukuri N, Belzile E. Does delirium increase hospital stay? J Am Geriatr Soc. 2003 Nov;51(11):1539-46. doi: 10.1046/j.1532-5415.2003.51509.x. PMID 14687382
- [Background] Inouye SK, Rushing JT, Foreman MD, Palmer RM, Pompei P. Does delirium contribute to poor hospital outcomes? A three-site epidemiologic study. J Gen Intern Med. 1998 Apr;13(4):234-42. doi: 10.1046/j.1525-1497.1998.00073.x. PMID 9565386
- [Background] Krogseth M, Wyller TB, Engedal K, Juliebo V. Delirium is a risk factor for institutionalization and functional decline in older hip fracture patients. J Psychosom Res. 2014 Jan;76(1):68-74. doi: 10.1016/j.jpsychores.2013.10.006. Epub 2013 Oct 16. PMID 24360144
- [Background] Leslie DL, Zhang Y, Holford TR, Bogardus ST, Leo-Summers LS, Inouye SK. Premature death associated with delirium at 1-year follow-up. Arch Intern Med. 2005 Jul 25;165(14):1657-62. doi: 10.1001/archinte.165.14.1657. PMID 16043686
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Background] Lopez S, Gros T, Bernard N, Plasse C, Capdevila X. Fascia iliaca compartment block for femoral bone fractures in prehospital care. Reg Anesth Pain Med. 2003 May-Jun;28(3):203-7. doi: 10.1053/rapm.2003.50134. PMID 12772137
- [Background] Dochez E, van Geffen GJ, Bruhn J, Hoogerwerf N, van de Pas H, Scheffer G. Prehospital administered fascia iliaca compartment block by emergency medical service nurses, a feasibility study. Scand J Trauma Resusc Emerg Med. 2014 Jun 23;22:38. doi: 10.1186/1757-7241-22-38. PMID 24957807
- [Background] Godoy Monzon D, Iserson KV, Vazquez JA. Single fascia iliaca compartment block for post-hip fracture pain relief. J Emerg Med. 2007 Apr;32(3):257-62. doi: 10.1016/j.jemermed.2006.08.011. Epub 2007 Feb 8. PMID 17394987
- [Background] Hogh A, Dremstrup L, Jensen SS, Lindholt J. Fascia iliaca compartment block performed by junior registrars as a supplement to pre-operative analgesia for patients with hip fracture. Strategies Trauma Limb Reconstr. 2008 Sep;3(2):65-70. doi: 10.1007/s11751-008-0037-9. Epub 2008 Sep 2. PMID 18762870
- [Background] Haines L, Dickman E, Ayvazyan S, Pearl M, Wu S, Rosenblum D, Likourezos A. Ultrasound-guided fascia iliaca compartment block for hip fractures in the emergency department. J Emerg Med. 2012 Oct;43(4):692-7. doi: 10.1016/j.jemermed.2012.01.050. Epub 2012 Apr 9. PMID 22494596
- [Background] Lees D, Harrison WD, Ankers T, A'Court J, Marriott A, Shipsey D, Chaplin A, Reed MR. Fascia iliaca compartment block for hip fractures: experience of integrating a new protocol across two hospital sites. Eur J Emerg Med. 2016 Feb;23(1):12-8. doi: 10.1097/MEJ.0000000000000167. PMID 24949565
- [Background] Hanna L, Gulati A, Graham A. The role of fascia iliaca blocks in hip fractures: a prospective case-control study and feasibility assessment of a junior-doctor-delivered service. ISRN Orthop. 2014 Mar 4;2014:191306. doi: 10.1155/2014/191306. eCollection 2014. PMID 24977087
- [Background] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- [Background] Adunsky A, Levy R, Heim M, Mizrahi E, Arad M. Meperidine analgesia and delirium in aged hip fracture patients. Arch Gerontol Geriatr. 2002 Nov-Dec;35(3):253-9. doi: 10.1016/s0167-4943(02)00045-6. PMID 14764364
- [Background] Candal-Couto JJ, McVie JL, Haslam N, Innes AR, Rushmer J. Pre-operative analgesia for patients with femoral neck fractures using a modified fascia iliaca block technique. Injury. 2005 Apr;36(4):505-10. doi: 10.1016/j.injury.2004.10.015. PMID 15755432
- [Background] Dulaney-Cripe E, Hadaway S, Bauman R, Trame C, Smith C, Sillaman B, Laughlin R. A continuous infusion fascia iliaca compartment block in hip fracture patients: a pilot study. J Clin Med Res. 2012 Feb;4(1):45-8. doi: 10.4021/jocmr724w. Epub 2012 Jan 17. PMID 22383926
- [Background] Cole MG. Delirium in elderly patients. Am J Geriatr Psychiatry. 2004 Jan-Feb;12(1):7-21. PMID 14729554
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- See also: European Union Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-003650-40/NL